CLINICAL TRIAL: NCT06262763
Title: Effect of High Intensity Laser on Sacroiliac Joint Pain In Adult Women
Brief Title: High-intensity Laser Therapy for Sacroiliac Joint Pain
Acronym: Girls
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Takwa Mohamed Saied Gado, Principle investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HILT for SIJP
Record Dates: First submitted 2024-02-06; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Sacroiliac Joint Pain
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Experimental): Laser with traditional exercises
  Interventions: Device: Laser Therapy; Other: Traditional exercises
- Group (B) (Placebo Comparator): Placebo LASER with traditional exercises
  Interventions: Other: Traditional exercises; Other: Placebo laser

INTERVENTIONS:
Device: Laser Therapy — High-intensity
  Other Names: High power
  Arms: Group (A)
Other: Traditional exercises — Hamstring and piriformis stretch, plank exercises and bird dog exercise
Other: Placebo laser — Not directed radiation to participant
  Arms: Group (B)

SUMMARY:
Effect of high intensity laser on sacroiliac joint pain

DETAILED DESCRIPTION:
Effect of high laser in reduction of pain and improve functional disability in adult women

ELIGIBILITY:
Inclusion Criteria:

* The presence of Pain over the sacroiliac joint with no surgical history.
* Unmarried.
* Tender SIJ on palpation.
* Workers with an average age of 18-30 years.
* Body mass index did not exceed 30 kg/m2.

Exclusion Criteria:

* If they have Infections. .Fracture in and around the SIJ Complex.
* Arthritis of joint.
* Pregnancy. .Smoking girls. .Patient not willing to participate in the study. .Any history of surgery. Lumbar spine disc herniation or back injury. Tumor around the joint.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2024-03-28 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | At the beginning and at after 12 session (1 month)
  By Visual Analogue Sclae (VAS)

SECONDARY OUTCOMES:
Pressure pain threshold | At the beginning and at after 12 session (1 month)
  By pressure algometer

OTHER OUTCOMES:
Functional disability | At the beginning and at after 12 session (1 month)
  By Oswestry index (Arabic version)

CONTACTS AND LOCATIONS:
Locations (1):
- Kafr Al-Sheikh University, Kafr ash Shaykh, Egypt